CLINICAL TRIAL: NCT05298969
Title: The Efficacy of Temporalis Myofascial Flap in Reconstruction of Various Cranio-maxillofacial Defects
Brief Title: Temporalis Myofascial Flap Effectiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Youssef Asham Gendy, Assistant Lecturer of ENT, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU 7
Record Dates: First submitted 2022-03-07; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Maxillary Sinus Neoplasms
Keywords: Temporalis flap; Maxillofacial defects; Reconstruction
MeSH Terms: conditions — Maxillary Sinus Neoplasms

STUDY DESIGN:
Intervention Model Description: Assessment of temporalis myofascial flap effectiveness in reconstruction of cranio-maxillofacial defects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flap survival (Experimental): Harvesting temporalis myofascial flap for cranio-maxillofacial defects
  Interventions: Procedure: Temporalis Myofascial flap

INTERVENTIONS:
Procedure: Temporalis Myofascial flap — Improvement of speech and feeding quality in patients with palatal defects by temporalis myofascial flap

SUMMARY:
This research is conducted as trial to improve lifestyle of patients with cranio-maxillofacial defects following major insults like trauma or tumor resection in form of speech problems or dysphagia by usage temporalis myofascial flap and assessment of it's effectiveness

ELIGIBILITY:
Inclusion Criteria:

* patients with:

  * TMJ ankylosis

    * Osteomyelitis following mucormycosis
    * Following tumor resection like maxillectomy or temporal bone resection
    * Following orbital exentration due to tumors or infections
    * Following massive trauma
    * Facial reanimation

Exclusion Criteria:

* • History of head & neck embolization as it may compromise blood supply of the flap

  * Extensive tumors involving maxillary artery
  * History of head & neck radiation or chemotherapy
  * Temporalis muscle wasting due to any reason
  * Bad general condition

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of versatility of temporalis myofascial flap in reconstruction of craniomaxillofacial defects in means of flap viability, healing and epithelization | 6 months postoperatively
  Assessment by regular follow up by pin bricks

SECONDARY OUTCOMES:
Assessment of phonation and swallowing efficacy postoperatively | 6 months postoperatively
  Assessment will be done in regular follow up visits by video fluoroscopy , trials of swallowing and phonation will be assessed by phoniatricians

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU7, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No